CLINICAL TRIAL: NCT02827331
Title: Taking Account of Inobservable Periods in Longitudinal Drug Treatment Follow-up
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31-14-7439
Record Dates: First submitted 2016-07-06; First posted 2016-07-11 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Drug Exposition
Keywords: Benzodiazepines; Fracture
MeSH Terms: conditions — Fractures, Bone | interventions — Hypnotics and Sedatives; Anti-Anxiety Agents; Prescriptions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Patients exposed to benzodiazepines: Data to be collected are :
  * Administrative and medical data
  * Exposition to hypnotics or anxiolytics benzodiazepines
  Interventions: Other: Exposition to hypnotics or anxiolytics benzodiazepines; Other: Administrative and medical data
- Patients not exposed to benzodiazepines: Data to be collected are :
  * Administrative and medical data
  * Exposition to non benzodiazepines antidepressants, hypnotics or anxiolytics
  Interventions: Other: Exposition to non benzodiazepines antidepressants, hypnotics or anxiolytics; Other: Administrative and medical data
- Control group: Data to be collected are :
  * Administrative and medical data
  * Medical consultation without prescription of interest
  Interventions: Other: Medical consultation without prescription; Other: Administrative and medical data

INTERVENTIONS:
Other: Exposition to hypnotics or anxiolytics benzodiazepines — Exposition to at least one drug belonging to the following classes during the last 12 months before index date :
  * Benzodiazepine derivatives (N05BA)
  * Benzodiazepine derivatives (N05CD)
  * Benzodiazepine related drugs (N05CF)
  Groups: Patients exposed to benzodiazepines
Other: Exposition to non benzodiazepines antidepressants, hypnotics or anxiolytics — Exposition to at least one drug belonging to the following classes during the last 12 months before index date :
  * Antipsychotics (N05A)
  * Antiepileptics with the exception of clonazepam (N03)
  * Drugs used for alcohol dependance (N07BB)
  * Drugs used for opioids dependance (N07BC)
  Groups: Patients not exposed to benzodiazepines
Other: Medical consultation without prescription — Medical consultation without prescription of any drugs of interest
  Groups: Control group
Other: Administrative and medical data — * Gender
  * Birthdate
  * Department of residence
  * City of residence
  * Vital status (month and date of death)
  * Affiliation to Universal Health Coverage
  * Number of chronic long-term illness, medical diagnostic or pathology (CIM 10 code), onset and end dates
  * Drugs reimbursements (Date of care onset, drugs identification code, number of box delivered)
  * Data collected from medicalisation program of information system and private and public home care structures
  * Medical consultations, medical acts ( Common Classification of Medical Acts nomenclature)

SUMMARY:
The question of the inclusion of periods of interruptions and periods unobservable has been studied as part of medico-administrative databases. However, the specificity of the health insurance databases justify the realization of dedicated methodological research. A thorough knowledge of the purpose of these data, how they collect and restitution is an essential prerequisite to carry out this work.

One type of scheme cohort exposed/unexposed led to the formulation of a finding on the basis of the comparison between the exposure groups. However, this traditional approach has the major drawback of neglecting the changing nature of drug exposure, and therefore fails to take into account any changes or interruptions doses. Approaches to take into account the time dependent variables were developed. These allow to take into account any interruptions. However, as part of study on health databases, sometimes we do not have the status in relation to the exhibition on the entire monitoring period. This is for example the case during hospitalization. The bias generated by the failure to take account of these periods ("non measurable time bias") can be problematic when a long exposure and chronic disorders require hospitalization.

ELIGIBILITY:
General Inclusion Criteria:

* Beneficiaries of all social security regimen with a minimum of one year of data in general sample of beneficiaries

Group expose to benzodiazepine :

* Exposition to at least one benzodiazepine or anxiolytic

Group antidepressants and anxiolytics and hypnotics non benzodiazepines :

* Exposition to at least one antidepressants and anxiolytics and hypnotics non benzodiazepines

Control group :

- Patient having a medical consultation without prescription of interest

Exclusion Criteria:

* Non incident patient : Patient having a prescription of benzodiazepines, clonazepam, tetrazepam, antidepressants, anxiolytics ou hypnotics non benzodiazepine during the last 12 months before index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population studied is from french general sample of beneficiaries. Patients are incident users of benzodiazepines
Sampling Method: Non-Probability Sample
Enrollment: 171861 (Actual)
Dates: Start 2014-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Comparison of mortality from all causes in the 3 groups as assessed by clinical data collected | through the end of study (12 months)
  Four approaches will be used :
  * intergroup comparison
  * Time influence with cox model
  * Use of markovian models
  * Inclusion of "non observable periods" with inobservable and observable death models

CONTACTS AND LOCATIONS:
Overall Officials: Maryse LAPEYRE-MESTRE, Study Director — University Hospital of Toulouse

IPD SHARING:
Plan to Share IPD: No